CLINICAL TRIAL: NCT04345276
Title: An Open Clinical Trial to Evaluate Danoprevir Sodium Tablets Combined With Ritonavir in the Treatment of SARS-CoV-2 Infection
Brief Title: Efficacy and Safety of Ganovo (Danoprevir) Combined With Ritonavir in the Treatment of SARS-CoV-2 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huoshenshan Hospital (Other)
Collaborators: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-CTP-HS-01
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Danoprevir+Ritonavir group (Experimental)
  Interventions: Drug: Danoprevir+Ritonavir

INTERVENTIONS:
Drug: Danoprevir+Ritonavir — Danoprevir 100mg , one tablet each time , twice per day, up to 10 days. Ritonavir 100mg, one tablet each time , twice per day, up to 10 days.
  Other Names: Ganovo

SUMMARY:
Evaluation of the efficacy and safety of Danoprevir sodium tablet combined with ritonavir for SARS-CoV-2 infected patients.

DETAILED DESCRIPTION:
Given no specific antiviral therapies for COVID-19 approved yet and Danoprevir sodium tablet, an oral Hepatitis C virus protease inhibitor, approved in China in June 2018 , this open, controlled trial will evaluate the efficacy and safety of Danoprevir sodium tablet in hospitalized patients infected with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old;
2. Pneumonia patients with SARS-CoV-2 infection were confirmed to be positive by RT-PCR and clinical manifestations. The diagnosis standard refers to the diagnosis and treatment plan for pneumonia with SARS-CoV-2 infection (Current Trial Version);
3. Patients with newly diagnosed respiratory system discomfort who have been hospitalized (the diagnosis time of respiratory system discomfort shall not exceed 7 days);
4. Women and their partners who have no planned pregnancy for nearly half a year and are willing to take effective contraceptive measures within 30 days from the first administration of the study drug to the last administration;
5. Agree not to participate in other clinical research within 30 days from the first administration of the study drug to the last administration;
6. Patients who voluntarily sign informed consent.

Exclusion Criteria:

1. The pneumonia patients with severe SARS-CoV-2 infection met one of the following conditions: respiratory distress, RR≥30 times / min; or SaO2 / SpO2≤93% in resting state; or arterial partial pressure of oxygen (PaO2) / concentration of oxygen (FiO2) ≤300MMHG (1mmhg = 0.133kpa);
2. Pneumonia patients with severe SARS-CoV-2 infection meet one of the following conditions: respiratory failure and need mechanical ventilation; or shock; or other organ failure combined with ICU monitoring treatment;
3. Severe liver disease (such as child Pugh score ≥C, AST > 5 times upper limit);
4. Patients with contraindications specified in the instructions of danoprevir and ritonavir tablets;
5. Patients who plan to take protease inhibitors other than danoprevir and ritonavir simultaneously during the trial.
6. The pregnancy test of female subjects in the screening period was positive;
7. The researchers judged that it was not suitable to participate in this clinical trial (for example, patients who may be transferred to another hospital during the study period; patients with multiple basic diseases, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of composite adverse outcomes | Within 10 days after administration
  Defined as SPO2≤ 93% without oxygen supplementation, PaO2/FiO2 ≤ 300mmHg or a respiratory rate ≥30 breaths per min without supplemental oxygen min without supplemental oxygen

SECONDARY OUTCOMES:
Time to recovery | Within 10 days after administration
  Clinical recovery was defined as sustained (48 hours) alleviation of illness based on symptom scores (fever, cough, diarrhea, myalgia, dyspnea) all being absent and no evidence for progression (newly-presented dyspnea, SpO2 decline ≥3%, respiratory rate ≥ 30 breaths per min without supplemental oxygen).
Rate of no fever | Within 10 days after administration
Rate of no cough | Within 10 days after administration
Rate of no dyspnea | Within 10 days after administration
Rate of no requiring supplemental oxygen | Within 10 days after administration
Rate of undetectable New coronavirus pathogen nucleic acid | Within 10 days after administration
Rate of mechanical ventilation | Within 10 days after administration
Rate of ICU admission | Within 10 days after administration
Rate of serious adverse event | Within 10 days after administration

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, MD, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- Huoshenshan Hostipal, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided